CLINICAL TRIAL: NCT06591195
Title: Distraction As Multimodal Pain Management for Children in Resource-constrained Settings (DISTRACT)
Brief Title: Distraction As Multimodal Pain Management
Acronym: DISTRACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BREC/00005194/2023
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Pain, Acute; Burns; Pediatric ALL
Keywords: Distraction; Pain treatment; Pediatric burn injury; Dressing change
MeSH Terms: conditions — Acute Pain; Burns; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Agnosia

STUDY DESIGN:
Intervention Model Description: Paediatric patients between the age of 5-12 years with minor and superficial partial thickness burn injuries who require dressing changes in the outpatient clinic, without sedation, will be randomized into two groups: the control group will receive standard practice of care which concerns a dressing change without any distraction methods, and the intervention group will receive distraction by use of a kaleidoscope as additional method for potential pain alleviation. Patients in both groups will receive paracetamol or non-steroidal anti-inflammatory drugs when required according to hospital protocol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking for allocation. After allocation, there is no possibility for blinding the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Distraction (Experimental): The intervention group will undergo a dressing change procedure with distraction by use of a kaleidoscope as additional method for pain alleviation. In both groups, patients will receive paracetamol or non-steroidal anti-inflammatory drugs when required according to hospital protocol.
  Interventions: Device: Distraction by use of kaleidoscope
- Control (No Intervention): The control group will undergo the standard dressing change procedure without additional distraction methods. In both groups, patients will receive paracetamol or non-steroidal anti-inflammatory drugs when required according to hospital protocol.

INTERVENTIONS:
Device: Distraction by use of kaleidoscope — À kaleidoscope is an optical device consisting of mirrors that reflect images of bits of coloured glass in a symmetrical geometric design through a viewer.
  A kaleidoscope was selected as the non-electronic method of distraction, because of its wide availability due to low costs, its evolving and colourful visual stimuli, the fact that is blocks out any visualisations from the environment when used properly, and because it requires active participation (i.e., greater attention) from the subject.
  Arms: Distraction

SUMMARY:
A randomized controlled trial will be performed at the Ngwelezana Hospital, Empangeni, South Africa. Paediatric patients between the age of 5-12 years with minor and superficial partial thickness burn injuries who require dressing changes in the outpatient clinic, without sedation, will be randomized into two groups: the control group will receive standard practice of care which concerns a dressing change without any distraction methods, and the intervention group will receive distraction by use of a kaleidoscope as additional method for potential pain alleviation. Patients in both groups will receive paracetamol or non-steroidal anti-inflammatory drugs when required according to hospital protocol. The primary outcome will be the change in pain score from pre-procedural to pain score during the dressing change and will be analysed with a linear regression analysis. Additionally, sub analyses will be performed to evaluate potentially modifying factors on the treatment effect. This will also be evaluated with a linear regression analysis. This will be correlated with care giver and health care worker observational pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between the age of 5 and 12 years old with burn injuries requiring dressing changes in the outpatient clinic, who in regular practice (non-research setting) would not receive any analgesics other than paracetamol or a non-steroidal anti-inflammatory drug (NSAID);
* Superficial partial thickness burns < 5% TBSA (total body surface area) at the time of injury
* Only the first change of dressing is included

Exclusion Criteria:

* Patients who underwent split skin grafts for their burns;
* Patients on sedatives or anti-epileptics;
* The use of pain-relieving medication other than paracetamol or NSAIDs;
* If it is the patient's second presentation to Ngwelezana hospital's outpatient burns department
* Painful additional injuries other than the burn injury;
* Physical or mental impairments which make it impossible to adequately comply with the trial protocol. For example, visual impairments, impaired ability to communicate, psychological comorbidities, and burns that limit the use of a kaleidoscope (facial burns or burns to both hands)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The difference in patient-reported pain score | Baseline, before wound cleaning (0 minutes) and after dressing change (within 10 minutes)
  The patient-reported pain score after the dressing change minus the pain score before the procedure. This pain score is rated on the Wong-Baker FACES Pain Rating Scale from 0-10.

SECONDARY OUTCOMES:
Observational pain score | During the dressing change procedure (0 minutes to 5 minutes)
  The observational pain score is measured during the dressing change on the Face, Legs, Activity, Cry and Consolability (FLACC) scale from 0 to 10. This score is corrected by the baseline (patiënt-reported) pain score before the dressing change.
Global satisfaction with treatment | After dressing change (within 10 minutes)
  Global satisfaction about the treatment is assessed among the patient's caregiver and healthcare provider. Global satisfaction will be rated on a 1-5 scale based on the question: "Considering pain relief, side effects, and emotional status, how satisfied were you with the dressing change your child underwent?"

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Naidoo, MD, Principal Investigator — General surgeon, head of Burns Unit at Ngwelezana Hospital, Empangeni, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haverkamp FJC, Naidoo R, Muhrbeck M, Pompermaier L, Wladis A, van Laarhoven CJHM, Tan ECTH. DISTRACT study: evaluating kaleidoscope distraction as part of multimodal pain management in paediatric dressing changes - study protocol of a single centre randomised trial. BMJ Open. 2025 Jul 28;15(7):e093761. doi: 10.1136/bmjopen-2024-093761. PMID 40721257